CLINICAL TRIAL: NCT03180554
Title: Body Versus Machine: Motivational Nondirective Resonance Breathing Versus Transcutaneous Vagus Nerve Stimulation in the Treatment of Fibromyalgia
Brief Title: Body Versus Machine: Deep Breathing Versus Vagus Stimulation for the Treatment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Ethan Paccione, M.S., M.A. (Other)
Responsible Party: Sponsor-Investigator, Charles Ethan Paccione, M.S., M.A., Ph.D. Fellow in Medicine and Health Sciences, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/8892; 2017046 (Other Grant/Funding Number: South-East Regional Health Authority)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Chronic Widespread Pain; Fibromyalgia
Keywords: chronic widespread pain; heart rate variability; pain intensity; diaphragmatic breathing; vagus nerve stimulation; fibromyalgia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Pain | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study will use a randomized controlled experimental design. A total of N=112 consenting CWP patients will be consecutively recruited from the Department of Pain Management and Research at Oslo University Hospital, Norway, and randomized to one of four intervention groups. Participants will be randomized to either a version 1 tVNS group, a version 2 tVNS group, a version 1 MNRB group, or a version 2 MNRB group. Both version 1 and 2 treatment interventions will be delivered at home, twice a day, for 15 min in the morning and for 15 min in the evening, for a total duration of 2 weeks. The participants' adherence to both interventions will be monitored electronically. An 80 % completion of tVNS stimulation and MNRB training will be regarded as adequate adherence in this project. Participants are invited to the clinic twice for pre- and post-intervention data collection.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All statistical analyses will be performed by a statistician who is blinded by participants' ID and health record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- tVNS version 1 (Other): Transcutaneous vagus nerve stimulation (tVNS) version 1 will be delivered non-invasively via a portable take-home stimulation device which attaches to the concha of the outer ear. Intensity, pulse duration, and frequency is optimised by the participant. Participants will receive a 15-minute stimulation twice a day (once in the morning upon waking and once in the evening before bed) for 2 weeks.
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)
- tVNS version 2 (Other): Transcutaneous vagus nerve stimulation (tVNS) version 2 will be delivered non-invasively via a portable take-home stimulation device which attaches to the center of the left ear lobe. Intensity, pulse duration, and frequency is optimised by the participant. Participants will receive a 15-minute stimulation twice a day (once in the morning upon waking and once in the evening before bed) for 2 weeks.
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)
- MNRB version 1 (Other): Motivational nondirective resonance breathing (MNRB) version 1 will be delivered via a take-home guided breathing apparatus. Participants will be guided through a deep breathing session. Participants will practice MNRB version 1 for 15-minutes twice a day (once in the morning upon waking and once in the evening before bed) for 2 weeks.
  Interventions: Other: Motivational nondirective resonance breathing (MNRB)
- MNRB version 2 (Other): Motivational nondirective resonance breathing (MNRB) version 2 will be delivered via a take-home guided breathing apparatus. Participants will be guided through a paced breathing session. Participants will practice MNRB version 2 for 15-minutes twice a day (once in the morning upon waking and once in the evening before bed) for 2 weeks.
  Interventions: Other: Motivational nondirective resonance breathing (MNRB)

INTERVENTIONS:
Device: Transcutaneous Vagal Nerve Stimulation (tVNS) — The tVNS system consists of a non-invasive, handheld stimulator and ear electrode that participants wear like an earphone. Intensity, pulse duration, and frequency of the tVNS stimulation is optimized in order to induce signals in thick-myelinated Aβ fibres of the auricular branch of the vagus nerve (ABVN).
  Other Names: Vagus Nerve Stimulation
  Arms: tVNS version 1; tVNS version 2
Other: Motivational nondirective resonance breathing (MNRB) — Motivational nondirective resonance breathing (MNRB) is a type of diaphragmatic breathing technique that trains the body to breathe at resonance frequency with a mental state of open-awareness.
  Other Names: Diaphragmatic Breathing
  Arms: MNRB version 1; MNRB version 2

SUMMARY:
This randomized controlled trial aims to compare the efficacy of two vagal nerve innervation treatments, motivational nondirective resonance breathing and transcutaneous vagus nerve stimulation, on heart rate variability and pain intensity in patients suffering from CWP. This project tests new and potentially effective means of treating a major global and public health concern where prevalence is high, disability is severe, and treatment options are limited.

DETAILED DESCRIPTION:
The primary objective of this randomized controlled trial is to investigate the effects of motivational nondirective resonance breathing (MNRB) and transcutaneous vagus nerve stimulation (tVNS) on autonomic health and pain intensity in participants diagnosed with chronic widespread pain (CWP). Two versions of MNRB and two versions of tVNS will be delivered and practiced by participants at home for two weeks. The primary outcome is photoplethysmography (PPG) measured heart rate variability (HRV). Secondary outcomes are self report numeric rating scale (NRS) pain intensity, FM pain severity and associated parameters, computerized cuff pressure algometry, blood pressure, psychological distress and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmatory diagnosis of chronic widespread pain, including fibromyalgia
* Widespread pain index (WPI) ≥ 7 and symptom severity scale (SSS) score ≥ 5 OR WPI of 4-6 and SSS score ≥ 9
* Generalized pain in at least 4 of 5 body regions must be present
* Pain symptoms have been generally present for at least 3 months
* Average pain intensity ≥ 6 on a 0-10 numerical rating scale, where 0 represents "no pain" and 10 represents the "worst pain imaginable"

Exclusion Criteria:

* History and/or presence of comorbid severe neurological or psychiatric disorders (e.g., mania, psychosis, suicidality, bipolar/schizophrenia/autism spectrum disorders)
* Neurodegenerative disorders (e.g., Parkinson´s, Alzheimer´s, Huntington´s disease)
* Pregnancy or planned pregnancy
* Planned surgery
* Eating disorder (e.g., obesity, anorexia nervosa, etc.)
* Head trauma
* Migraine
* Active heart implants (e.g., pacemaker)
* Active ear implants (e.g., cochlear implant)
* Individuals who have practiced meditation consistently (for more than 20 min/day) within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Heart Rate Variability (HRV) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  The root mean square of successive differences (RMSSD) will be derived from photoplethysmography (PPG) recordings and serve as the primary HRV outcome of interest. RMSSD corresponds to the parasympathetic regulation of heart beats (i.e. vagal activity) which is associated with self-report average pain intensity in CWP patients. Three readings on the right index finger are taken in a sitting position, separated by a one minute intervals, and after a five minute acclimatization (resting) period. The average of the last two measurements will be used in the final analyses.

SECONDARY OUTCOMES:
Change from Baseline Numeric Rating Scale (NRS) for Average Pain Intensity | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  The NRS for pain is a unidimensional measure of pain intensity in adults. It is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain where 0 represents ''no pain'' and 10 represents ''the worst pain imaginable''.
Change from Baseline Fibromyalgia severity (FS) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  FS is a self-report measure of a participant´s overall CWP/fibromyalgia severity composed of their widespread pain index (WPI) and symptom severity scale (SSS). The WPI (0-19) is the number of areas in which the patient has had pain over the last week (0-19). The SSS (0-12) is the sum of the severity scores of 3 symptoms (fatigue, waking unrefreshed, and cognitive symptoms) (0-9) plus the sum (0-3) of the number of the following symptoms the patient has been bothered by that occurred during the previous 6 months: (1) Headaches (0-1) (2) Pain or cramps in lower abdomen (0-1) (3) And depression (0-1). The fibromyalgia severity (FS) scale is the sum of the WPI and SSS.
Change from Baseline Pain Detection Threshold (PDT), Pain Tolerance Threshold (PTT), and Pressure-Pain Limit (PPL) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  Computerized cuff pressure algometry (CPA) will be used in order to safely and efficiently assess pain sensitivity mechanisms in CWP patients. The cuff will be placed on the mid-portion of the dominant lower leg and will use ramp inflation of 1 kPa/s until subjects indicate PDT, PTT, and PPL which is based upon an electronic 10cm visual analogue scale (VAS). PDT is the pressure value at the moment of transition between strong and painful pressure (the first time the VAS exceeds 0) whereas PTT is defined as the pressure value at the termination of pressure inflation (the corresponding VAS score is the PPL). The zero and 10 cm extremes on the VAS are defined accordingly as ''no pain'' and as ''the worst pain imaginable''.The subject is instructed to rate the pain intensity continuously on the VAS from the first sensation of pain and to press the hand-held pressure release button when the pain becomes unbearable. An average of three recordings will be used in the final analyses.
The Hopkins Symptom Checklist-25 (HSCL-25) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  The HSCL-25 assesses emotional distress, anxiety, and depressive symptoms. The HSCL-25 scale consists of 25 questions about the presence and intensity of the most common psychiatric symptoms of anxiety and depression. Participants are asked: "To what extent have you been bothered by the following symptoms in the last 14 days including today?" Responses include: 1 (not at all), 2 (a little), 3 (quite a bit) and 4 (extremely).
Change from Baseline Blood Pressure (BP) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  Resting systolic and diastolic BP will be measured using an automated oscillometric device. The correct size cuff is chosen after the circumference of the upper arm is measured. Following a two minute rest, three readings on the upper right arm are taken in a sitting position separated by one minute intervals. The average of the last two readings will be used in the final analyses.
EQ-5D-5L | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  The EQ-5D-5L is a standardized instrument to measure health-related quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of these dimensions has 5 levels: "no problems," "slight problems," "moderate problems," "severe problems" and "extreme problems". The digits for the five dimensions are then combined into a 5-digit number that describes the patient's health state. The EQ VAS uses a vertical visual analogue scale from 0 - 100 to record the patient's current state of health. The endpoints on the EQ VAS are labelled 'The best health you can imagine', indicated by 100, and 'The worst health you can imagine', indicated by 0.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  The MAIA assesses participants' interoceptive body awareness and provides pertinent information in regards to how emotions and the perception of pain are related to interoception. The MAIA is a 32-item multidimensional instrument comprising of eight scales (e.g. noticing, non-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting) ranging from 3 to 7 items each. Each of the 32-items are scored from a 0 to a 5 which indicates how often each statement applies in daily life (where 0 represents "never" and a 5 represents "always"). The average of all eight scales is then computed as a final score.
Spirituality and Coping (SpREUK-15) | Baseline (Pre-2 week Intervention); Post-2 week Intervention
  The SpREUK-15 investigates whether or not participants rely on spirituality as a resource to cope with pain. It investigates three factors: 1) having trust/faith; 2) search for a transcendent source to rely on; and 3) reflection of life and subsequent change of life and behavior. Items are scored on a 5-point scale from disagreement to agreement (0 - does not apply at all; 1 - does not truly apply; 2 - don't know (neither yes nor no); 3 - applies quite a bit; 4 - applies very much). The scores can be referred to a 100% level (transformed scale score). Scores > 50% indicate higher agreement (positive attitude), while scores < 50 indicate disagreement (negative attitude).
Patient Global Impression of Change (PGIC) | Post-2 week Intervention
  The PGIC is a self-report measure of participant belief about the efficacy of a treatment and their overall improvement. Participants rate their change on a 7 point scale: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse".
Credibility / Expectancy Questionnaire (CEQ) | Baseline (Pre-2 week Intervention)
  The CEQ is a a self-report measure of a participant´s expectations about the efficacy of a particular treatment and whether they think that the treatment is credible or not. In particular, it investigates two factors-- what one feels and what one thinks in regards to the treatment. The CEQ is composed of six items which are scored on a 9 point scale ranging from: "not at all logical", "somewhat logical", and "very logical". Items 4 and 6 ask the participant how they feel and how they think the administered treatment will improve their overall health state in regards to their pain on a 0 - 100% scale, where 0% represents "no improvement" whereas 100% represents "total improvement".

CONTACTS AND LOCATIONS:
Overall Officials: Audun Stubhaug, M.D., D.Med.Sci., Study Director — Oslo University Hospital; Leiv Arne Rosseland, M.D.,Ph.D., Study Chair — Oslo University Hospital; Henrik B Jacobsen, Ph.D., Principal Investigator — Oslo University Hospital; Charles E Paccione, M.S., M.A., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Department of Pain Management and Research, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
All data will be de-identified. Data points will be reduced to ensure anonymity and will be uploaded to a server yet to be determined.

REFERENCES:
- [Derived] Paccione CE, Stubhaug A, Diep LM, Rosseland LA, Jacobsen HB. Meditative-based diaphragmatic breathing vs. vagus nerve stimulation in the treatment of fibromyalgia-A randomized controlled trial: Body vs. machine. Front Neurol. 2022 Nov 3;13:1030927. doi: 10.3389/fneur.2022.1030927. eCollection 2022. PMID 36438970
- [Derived] Paccione CE, Diep LM, Stubhaug A, Jacobsen HB. Motivational nondirective resonance breathing versus transcutaneous vagus nerve stimulation in the treatment of fibromyalgia: study protocol for a randomized controlled trial. Trials. 2020 Sep 23;21(1):808. doi: 10.1186/s13063-020-04703-6. PMID 32967704